CLINICAL TRIAL: NCT05944952
Title: A Pilot Study Comparing a Low-dose Versus a High-dose Sublingual Buprenorphine Induction Dosing Scheme in Fentanyl Using Patients With Opioid Use Disorder (OUD)
Brief Title: Low-dose Versus a High-dose Sublingual Buprenorphine Induction
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: MATClinics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either the low-dose (n=20) or high dose (n=20) group and dispensed medication daily for one week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- high dose (Experimental): High dose: Participants randomized to the high dose group will receive on day 1 in the clinic an initial dose of 2 mg of buprenorphine/naloxone, followed by a 6 mg dose an hour later, followed by an 8 mg dose an hour later, followed by an 8 mg dose an hour later. On day 2 they will receive a 12 mg dose in the clinic and a 12 mg dose as take-home medication. On days 3 through 7 they will report to the clinic and receive their 12 mg morning dose and a 12 mg dose as a take-home for evening dosing. Thereafter, dosing adjustments can be made in the first three months of the trial.
  Interventions: Drug: buprenorphine/naloxone
- low dose (Active Comparator): Low dose: Participants randomized to the low dose group will receive 0.5 mg of buprenorphine/naloxone on day 1, 0.5 mg bid on day 2, 1.0 mg bid on day 3, 2.0 mg bid on day 4, 4.0 mg bid on day 5, 4.0 mg tid on day 6, and 8 mg bid on day 7. Thereafter, dosing adjustments can be made in the first three months of the trial.
  Interventions: Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: buprenorphine/naloxone — Participants will be dosed with buprenorphine/ naloxone strips
  Other Names: suboxone

SUMMARY:
This study proposes to compare a low-dose versus a high-dose buprenorphine induction scheme in 40 fentanyl using people with Opioid Use Disorder (OUD). Study participants will be randomized to either the low-dose (n=20) or high dose (n=20) group and dispensed medication daily for one week.

DETAILED DESCRIPTION:
This study proposes to compare a low-dose versus a high-dose buprenorphine induction scheme in 40 fentanyl using people with Opioid Use Disorder (OUD). Study participants will be randomized to either the low-dose (n=20) or high dose (n=20) group and dispensed medication daily for one week. Thereafter, they will be treated according to the MATClinics usual schedule of clinic visits. The number and timing of visits may vary according to whether the participant is still using illicit opioids. Follow-up visits for the study will be at one and three months.The primary objective is to determine whether patients randomly assigned to low versus high dose induction regimens are more likely to complete the 7-day induction period. Secondary outcomes are the number of patients who develop precipitated withdrawal or other adverse events, experience subjective opioid withdrawal symptoms, use adjunctive medications (hydroxyzine, loperamide, dicyclomine, clonidine, ibuprofen, methocarbamol, trazodone, ondansetron) provided by the clinic, recommendation of the medication induction scheme to other patients, and treatment retention at 1- and 3- months post induction.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (≥ 18 years of age) persons with a DSM-5 diagnosis of OUD;
* Must have a fentanyl positive urine test;
* Able to come to the clinic every day for the first week of treatment.

Exclusion Criteria:

* No exclusionary medical history or mental health issues as determined by the admitting provider; e.g., patients with untreated or unstable serious mental illness, including psychotic disorders;
* Alcohol withdrawal requiring pharmacological management;
* Urine positive for buprenorphine, benzodiazepines, or methadone; 4. Enrolled in a methadone treatment program in the past 14 days; 5. Inability to pass a study enrollment quiz.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
pharmacotherapy adherence | 1-7 days
  completion of dose induction regimen (yes/no)
pharmacotherapy adherence | out of 7 days
  number of days adherent to dose induction regiment

SECONDARY OUTCOMES:
Clinical Opiate Withdrawl Scale (COWS) | 1-7 days
  Precipitated withdrawal symptoms score; 11-item scale Score: 5- 12 = mild; 1 3-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal
Illicit opioid urine test results | baseline, 1-7 days, 1 month, 3month
  Positive opioid urine drug screen
Time Line Follow-Back (TLFB) Self-reported illicit opioid use | baseline, 1-7 days, 1 month, 3 month
  Self-report daily during first week then number of days during the past 30 for 1 and 3 month follow-ups
Subjective Opiate Withdrawal Scale (SOWS) | 1-7 days
  Subjective opioid withdrawal symptoms score (1-10, mild withdrawal; 11-20 moderate withdrawal; 21-30 severe withdrawal)
Adjunctive medications | 1-7 days
  Use of any adjunctive meds by self-report
Concomitant medications checklist | 1-7 days, 1 month, 3 month
  Any medication taken by the participant to treat a medical or psychiatric disorder
Adverse events (AEs) reporting form | baseline, 1-7 days, 1 month, 3 month
  Any reaction, side effect, or untoward event that occurs during the clinical trial, including reported overdoses

CONTACTS AND LOCATIONS:
Locations (1):
- MATClinics, Dundalk, Maryland, United States